# **Statistical Analysis Plan**

Bioequivalence ProtocolPPDProject Code: PPDIdentification No.Merck Protocol Number: MS200084 0015

**Title:** A randomized, open-label, two-way crossover study assessing

the bioequivalence (BE) between single dose of 750 mg Glucophage® XR Tablets (PT Merck Tbk, Jakarta, Indonesia-Manufactured) and 750 mg Glucophage® XR Tablets (Merck Santé, Semoy, France-Manufactured) under fasted state in

healthy subjects

**Study Phase** Phase I (Bioequivalence Study)

**Investigational Medicinal** Glucophage XR® 750 mg

Product(s)

**Clinical Study Protocol** 

Version

Version 1.1, 22-May-2018

Statistical Analysis Plan PPD

**Author** 

Statistical Analysis Plan Version 1.0, 06-Sep-2018

Date and Version

Statistical Analysis Plan

Reviewers

PPD ,PPD

PPD , Clinical Pharmacologist

PPD , Clinical Pharmacologist

PPD , Local Medical Responsible

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies.

It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2018 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

# 1 Signature Page

## Statistical Analysis Plan: MS200084\_0015

A randomized, open-label, two-way crossover study assessing the bioequivalence (BE) between single dose of 750 mg Glucophage® XR Tablets (PT Merck Tbk, Jakarta, Indonesia-Manufactured) and 750 mg Glucophage® XR Tablets (Merck Santé, Semoy, France-Manufactured) under fasted state in healthy subjects

| Statistical Apalysis Plan Author: | |
|----------------------------------------------|-------|
| PD | |
| | PPD |
| | Date |
| Charles I A a levie Dlan American | |
| Statistical Analysis Plan Approver: | |
| | PPD |
| | r r D |
| PPD | Date |
| PPD / Local Medical Responsible | Bate |
| PT Merck Tbk | |
| Perkantoran Hijau Arkadia F Tower 15th Floor | |
| Jl. TB Simatupang Kav 88, Pasar Minggu | |
| Jakarta 12520 – INDONESIA | |

| 2 | Table of Contents | |
|--------|----------------------------------------------------------------|----|
| 1 | Signature Page | 2 |
| 2 | Table of Contents | 3 |
| 3 | List of Abbreviations and Definition of Terms | 5 |
| 4 | Modification History | 8 |
| 5 | Purpose of the Statistical Analysis Plan | 8 |
| 6 | Summary of Clinical Study Features | 8 |
| 7 | Sample Size/Randomization | 12 |
| 8 | Overview of Planned Analyses | 13 |
| 9 | Changes to the Planned Analyses in the Clinical Study Protocol | 13 |
| 10 | Protocol Deviations and Analysis Sets | 14 |
| 10.1 | Definition of Protocol Deviations and Analysis Sets | 14 |
| 10.2 | Definition of Analysis Sets and Subgroups | 14 |
| 11 | General Specifications for Statistical Analyses | 14 |
| 12 | Study Subjects | 15 |
| 12.1 | Disposition of Subjects and Discontinuations | 15 |
| 12.2 | Protocol Deviations | 16 |
| 12.2.1 | Important Protocol Deviations | 16 |
| 12.2.2 | Reasons Leading to the Exclusion from an Analysis Set | 16 |
| 13 | Demographics and Other Baseline Characteristics | 16 |
| 13.1 | Demographics | 16 |
| 13.2 | Medical History | 17 |
| 13.3 | Other Baseline Characteristics | 17 |
| 14 | Previous or Concomitant Medications/Procedures | 18 |
| 15 | Treatment Compliance and Exposure | 19 |
| 16 | Endpoint Evaluation | 19 |
| 16.1 | Primary Endpoint Analyses | 19 |
| 16.2 | Secondary Endpoint Analyses | 19 |
| 16.3 | Estimation of Individual PK Parameters | 20 |
| 17 | Safety Evaluation | 20 |
| 17.1 | Adverse Events | 20 |

| 17.1.1 | All Adverse Events | 21 |
|---|---|---|
| 17.1.2 | Adverse Events Leading to Treatment Discontinuation | 23 |
| 17.2 | Deaths, Other Serious Adverse Events, and Other Significant Adverse Even | nts24 |
| 17.2.1 | Deaths | 24 |
| 17.2.2 | Serious Adverse Events | 24 |
| 17.3 | Clinical Laboratory Evaluation | 24 |
| 17.4 | Vital Signs | 26 |
| 17.5 | Other Safety or Tolerability Evaluations | 26 |
| 18 | Benefit Risk Assessment | 27 |
| 19 | References | 27 |
| List of Tabl | es | |
| Table 1 | Demographic Data | 16 |
| Table 2 | Clinical Laboratory Test and ECG of Subjects | 17 |
| Table 3 | List of Adverse Events Occurred | 22 |
| Table 4 | Overview of all Adverse Events (by Group and Overall) | 22 |
| Table 5 | Adverse Events: Number Observed | 23 |
| Table 6 | Listing of Subjects Who Dropped Out from Study | 23 |
| Table 7 | Listing of Deaths During the Study | 24 |
| Table 8 | Listing of Serious Adverse Events | 24 |
| Table 9 | Clinical Laboratory Test and ECG of Subjects During Follow-Up Visit | 25 |
| Table 10 | Vital Signs Monitoring | 26 |
| Table 11 | Unscheduled Measurement | 26 |

## 3 List of Abbreviations and Definition of Terms

μL Microlitre

AE Adverse Event

ALT Alanine minotransferase
ANOVA Analysis of Variance
AP Alkaline Phosphatase

ASEAN Association of Southeast Asian Nations

AST Aspartate aminotransferase

AUC<sub>0-inf</sub> Area under plasma concentration versus time curve extrapolated to infinite time

AUC<sub>0-t</sub> Area under plasma concentration versus time curve from administration to last

observed concentration at time t

BPOM Badan Pengawasan Obat dan Makanan (the Indonesian National Agency of

Drug and Food Control, NA-DFC)

BE Bioequivalence
BMI Body mass index
BP Blood pressure

BQL Below the quantification limit

CI Confidence interval

C<sub>max</sub> Maximum observed plasma concentration

CRF Case Report Form

CV Coefficient of variation
CSR Clinical Study Report

dL Decilitre

ECG Electrocardiogram

EMA European Medicines Agency

EU Ehrlich units (corresponding to one milligram of urobilinogen per deciliter of

sample)

F Female

FDA Food and Drug Administration

FU Follow-up

g Gram

GCP Good Clinical Practice

h Hour

Hb Hemoglobin

HBsAg Hepatitis B Surface Antigen

HCG Human chorionic gonadotropin

HCV Hepatitis C Virus

HIV Human Immunodeficiency Virus

HPF High Power Field

HPLC-UV High Performance Liquid Chromatography with Ultraviolet Detector

ICH International Conference on Harmonization

ID Identification

IU International Unit

kg Kilogram

L Litre

ln Natural logarithm

M Male m Metre

Max Maximum

Mean Arithmetic mean

mg Milligram
ms Milliseconds
Min Minimum
min Minute(s)
mL Millilitre

mmHg Millimetre mercury column

N Number of non-missing observations

Neg. Negative

PK Pharmacokinetics

Pos. Positive

QTc Corrected QT interval

R Comparator drug

RBC Red Blood Cells

SAE Serious Adverse Event
SAP Statistical Analysis Plan

SD Standard DeviationSOC System Organ Class

T Test drug

 $t_{1/2}$  Elimination half-life

t<sub>max</sub> Time to reach maximum plasma concentration

ULN Upper limit of normal WBC White Blood Cells

WHO-ART World Health Organization Adverse Reaction Terminology

WOCBP Women of childbearing potential

XR Extended Release

yr Year

# **4 Modification History**

| Unique<br>Identifier for<br>SAP Version | Date of<br>SAP Version | Author | Changes from the Previous Version |
|---|---|---|---|
| 1.0 | 06-Sep-2018 | PPD | Not applicable |

# 5 Purpose of the Statistical Analysis Plan

The purpose of this SAP is to document technical and detailed specifications for the final analysis of data collected for study protocol MS200084\_0015. Results of the analyses described in this SAP will be included in the Clinical Study Report (CSR). Any post-hoc, or unplanned analyses performed to provide results for inclusion in the CSR but not identified in this prospective SAP will be clearly identified in the CSR.

The SAP is based upon the study protocol (version 1.1 dated 22 May 2018) and is prepared in compliance with ICH E9.

# **6** Summary of Clinical Study Features

#### **Objective**

Primary objective:

• To assess bioequivalence between metformin hydrochloride (Glucophage® XR) manufactured in PT Merck Tbk, Indonesia (test drug) and metformin hydrochloride (Glucophage® XR) manufactured in Merck Sante, France (comparator drug) following single oral dose administration under fasting condition.

#### Secondary objective:

- To compare pharmacokinetic parameters of metformin after single dose administrations of test and comparator (reference) drugs.
- To examine the safety and tolerability of metformin after single dose administrations of test and comparator (reference) drugs.

#### **Study Design**

An open-label, randomized, single-dose, two-period, two-sequence crossover study under fasting conditions

#### **Study Subjects**

Forty-eight (48) healthy adult male and female subjects



#### **Dosing Regimen**

- One (1) Glucophage® XR 750 mg Tablet produced by PT Merck Tbk, Indonesia of test drug (T) given as a single oral dose with approximately 200 mL of water at ambient temperature after an overnight fast of at least 10 hours.
- One (1) Glucophage® XR 750 mg Tablet produced by Merck Sante, France of comparator drug (R) given as a single oral dose with approximately 200 mL of water at ambient temperature after an overnight fast of at least 10 hours.

#### Washout

At least 7 days between doses.

#### **Duration of the Clinical Phase**

The duration of the clinical phase (from Screening through Follow-Up Study) will be approximately 6 weeks.

#### **Inclusion criteria**:

- Subject has provided written informed consent prior to the conduct of any study-related activities.
- Male and female subjects.
- Aged between 18 and 55 years, inclusive.
- Body mass index of 18 to 25 kg/m<sup>2</sup>.
- Good physical and mental health status, determined on the basis of medical history and physical examination.
- Vital signs (blood pressure, pulse rate, respiratory rate and body temperature) in sitting position within the normal range or showing no clinically relevant deviation per the Investigator's opinion.
- All values for laboratory assessments (hematology, clinical chemistry and urinalysis) within the normal range or showing no clinically relevant deviation per the Investigator's opinion.
- No clinically significant abnormality on 12-lead electrocardiogram (ECG) recording as judged by the Investigator; QTc (Bazett) should be  $\leq 450$ ms.
- Non-smoker or smoker less than 10 cigarettes per day.
- Women of childbearing potential (WOCBP) who are not nursing, are not pregnant, and are using highly effective methods of birth control (defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1 percent per year) when used consistently and correctly) for a period of at least one month before and after dosing. Standard birth control methods are considered to be: oral or implanted contraceptive therapy and intra-uterine devices. Female subjects may also be enrolled if they are postmenopausal (i.e., at least

12 consecutive months of amenorrhea after the last menstrual period) or surgically sterilized/hysterectomized at least 6 months prior to study participation.

- WOCBP must have a negative urine pregnancy test at Screening and on each admission (Day 1 of each dosing period).
- Negative screen for alcohol and drugs abuse (opiate class, barbiturates, cocaine and metabolites, amphetamines, cannabinoids and benzodiazepines) at Screening and on each admission (Day 1 of each dosing period).
- Negative screen for Hepatitis B surface antigen (HBsAg), HCV antibodies and/or HIV antibodies.

#### **Exclusion criteria**:

- Participation in a clinical study within 90 days prior to Screening.
- Blood donation (equal or more than 300 mL) or significant blood loss within 90 days prior to first drug administration.
- Any surgical or medical condition, including findings in the medical history or in the prestudy assessments, or any other significant disease, that in the opinion of the investigator, constitutes a risk or a contraindication for the participation of the subject in the study or that could interfere with the study objectives, conduct or evaluation.
- History of malignant diseases, except in-situ basal cell skin tumors treated with curative intent.
- History of surgery of the gastrointestinal tract which could influence the gastrointestinal absorption and/or motility per the Investigator's opinion.
- History or presence of relevant liver diseases or hepatic dysfunction (laboratory result for liver function test ≥ 1.5 ULN).
- History or presence of renal failure or renal dysfunction based on clinical symptoms and finding (serum creatinine concentration >1.4 mg/mL).
- Ascertained or presumptive hypersensitivity to the active drug substance and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study.
- Receipt of any prescription or non-prescription medication within 14 days before the first drug administration, except for hormonal contraceptives in female, and including multivitamins and herbal products (e.g. St John's Wort).
- Consumption of large quantities of methylxanthine-containing beverages (> 5 cups of coffee/day or equivalent).
- Consumption of grapefruit, orange, cranberry or juices of these three fruits, 24 hours prior to drug administration.
- Known lack of subject compliance or inability to communicate or cooperate with the Investigator (e.g., language problem, poor mental status).

#### **Pharmacokinetic Sampling**

- Eighteen (18) blood samples (1 x 10 mL and 17 × 5 mL) per subject in each period for drug content analysis.
- A 10-mL blood sample (control) will be drawn from fasting subjects immediately before drug administration.
- Subsequent blood samples are drawn 5 mL each at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24, and 32 hours after drug administration.
- Subjects who complete both periods will have a total of 36 blood samples collected. Total blood volume collection is approximately 210 mL (including 10 mL for Screening, 10 mL for each pre-dose period, 85 mL during each dosing period, and 10 mL for Follow-Up Visit).

#### **Bioanalytical Sample Analyses**

The metformin plasma concentrations will be measured using a validated high-performance liquid chromatography with ultraviolet detection (HPLC-UV; Waters<sup>TM</sup>, PPD) and according to the bioanalytical laboratory's standard operating procedures and applicable regulatory requirements.

#### **Pharmacokinetic Parameters**

Pharmacokinetic parameters:  $AUC_{0-t}$ ,  $AUC_{0-inf}$ ,  $C_{max}$ ,  $t_{max}$ , and  $t_{1/2}$ 

#### **Statistical Methods**

- Pharmacokinetic analyses will be performed using standard non-compartmental methods of Phoenix<sup>®</sup> WinNonlin (PPD ).
- The statistical method for testing bioequivalence is ANOVA for two-period, two-sequence, two-treatment cross-over comparing AUC<sub>0-t</sub> and C<sub>max</sub> after ln transformation of the original values. The terms to be used in the ANOVA model are sequence, subject within sequence, period, and formulation. The t<sub>max</sub> are compared using non-parametric test from the original data. The difference in t<sub>max</sub> will be analyzed non-parametrically on the original data using Wilcoxon matched-pairs test. The t<sub>½</sub> difference will be analyzed using Student's paired t-test or Wilcoxon matched-pairs test depending whether the differences of the paired data were distributed normally or not.

#### **Bioequivalence Criteria**

Bioequivalence is concluded if the 90% confidence interval of the Test/Reference geometric means ratio is in the range of 80.00-125.00% for AUC<sub>0-t</sub> and C<sub>max</sub>. This acceptance criterion is according to the Guideline on the Investigation of Bioequivalence, EMA, London, 2010; ASEAN Guideline for the Conduct of Bioequivalence Study, Lao PDR, 2015; and *Indonesian guidelines, Pedoman Uji Bioekivalensi, Badan Pengawas Obat dan Makanan (BPOM), Jakarta, 2015, page 37-38*.

# 7 Sample Size/Randomization

The number of subjects needed for a bioequivalence study was calculated with the following equation:

$$N = \frac{2 \cdot s_w^2 \cdot (Z_{1-\beta} + Z_{1-\alpha})^2}{(Ln(\mu_T / \mu_R) - Ln(1.25))^2}$$
$$S_w^2 = Ln(1 + (CV)^2)$$

 $\alpha$ : significance level (5%)

 $\beta$ : power (20%)

 $\mu_T$  : average score of bioavailability parameters for the test drug

 $\mu_R$  : average score of bioavailability parameters for the comparator drug

CV : intra-subject CV

CCI

. If these CVs are applied together with applicable bioequivalence criteria for AUC and C<sub>max</sub> (0.80-1.25), and the true treatment ratio Test/Reference is allowed to vary within 0.95 and 1.05, then 44 evaluable subjects will provide at least 90% power to show bioequivalence. Per *Indonesian guidelines*, *Pedoman Uji Bioekivalensi*, *Badan Pengawas Obat dan Makanan (BPOM)*, *Jakarta*, 2015, page 20, only 80% power is required at the minimum.

For a compensation of possible drop-outs during the study, an additional four (4) subjects shall be included based on the site's standard practice. Subjects will not be replaced, even if there are more than four (4) drop-outs.

A total of forty-eight (48) healthy adult male and female subjects shall thus be included in this study with no reserve subjects. 48 subjects will be administered with the study drug and the blood will be taken at various time points of blood sampling procedures. The blood samples from 48 subjects will be analyzed for plasma concentrations of metformin.

#### **Randomization Sequence**

Sequence 1 = TR (24 subjects)

Sequence 2 = RT (24 subjects)

The randomization code is tabulated for all subjects according to block randomization with a block size of 4 (Dixon & Massey, 1969, page 449). Subjects will be randomly allocated to one of the 2 treatment sequences (TR or RT) based on their assigned subject number. The randomization to a treatment sequence will be performed before the first period of the study.

Each study drug (test and reference drug) will be placed in a sealed envelope indicated with the subject number and its intended period and segregated in different labeled boxes kept in a limited access drug storage room. The study drugs will be dispensed to the study subjects by an

unblinded pharmacist prior to time of dosing. The randomization will be balanced according to subject number and the randomization code will be kept under controlled access. The clinical personnel administering the study drugs and the subjects are not blinded. The randomization code will not be available to the bioanalytical personnel (blinded for bioanalytical facility) till code breaking.

Code breaking will be performed after database lock i.e. after analysis of all blood samples has been finalized, and all PK parameters have been calculated. Sponsor's green light has to be obtained prior to code breaking, upon satisfying pre-defined conditions.

# 8 Overview of Planned Analyses

Pharmacokinetic and statistical analyses will be performed for metformin plasma data.

For pharmacokinetic calculations the actual sampling time will be used for any deviation in sample collection time (for post-dose blood sampling time points) from the scheduled time beyond the specified window period.

All concentration values below the quantification limit (BQL) will be set to zero for all pharmacokinetic and statistical calculations. However, it will be reported as BQL in the CSR (FDA, Bioanalytical Method Validation, May 2018, p.13).

If the pre-dose concentration is  $\leq$  5 percent of  $C_{max}$  value in that subject, the subject's data without any adjustments can be included in all pharmacokinetic measurements and calculations. If there are any subjects for whom the pre-dose concentration is > 5 percent of the  $C_{max}$  value for the subject in that period, the subject will be dropped from all BE study evaluations.

Pharmacokinetic analyses will be performed using standard non-compartmental methods of Phoenix® WinNonlin® (PPD ).

The statistical method for testing bioequivalence is ANOVA for 2-period, 2-sequence, 2-treatment cross-over comparing  $AUC_{0-t}$  and  $C_{max}$  after ln transformation of the original values. The  $t_{max}$  are compared using non-parametric test from the original data. The difference in  $t_{max}$  will be analyzed non-parametrically on the original data using Wilcoxon matched-pairs test. The  $t_{1/2}$  difference will be analyzed using Student's paired t-test or Wilcoxon matched-pairs test depending whether the differences of the paired data were distributed normally or not.

# 9 Changes to the Planned Analyses in the Clinical Study Protocol

The statistical methods as described in the protocol were adopted. There are no changes to the planned analyses.

# 10 Protocol Deviations and Analysis Sets

#### 10.1 Definition of Protocol Deviations

Important protocol deviations are protocol deviations that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a subject's rights, safety, or well-being.

Important protocol deviations include:

- Subjects that are dosed on the study despite not satisfying the inclusion criteria;
- Subjects that develop withdrawal criteria whilst on the study but are not withdrawn;
- Subjects that receive the wrong treatment or an incorrect dose;
- Subjects that receive an excluded concomitant medication;
- Deviations from scheduled sampling time points outside of the defined window period;
- Deviation from GCP.

# 10.2 Definition of Analysis Sets and Subgroups

#### Safety Analysis Set

The safety analysis will include all subjects who have received at least one dose of the investigational product and have had one subsequent safety assessment.

## **PK Analysis Set**

The PK analysis set will include all subjects without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results, with adequate trial medication compliance, and who have valid primary endpoints for both treatment.

# 11 General Specifications for Statistical Analyses

PK concentration data will be descriptively summarized using: number of non-missing observations (N), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), minimum (Min), median (Median) and maximum (Max).

PK parameter data will be descriptively summarized using: number of non-missing observations (N), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), minimum (Min), median (Median), maximum (Max), geometric mean, and the 90% confidence interval.

For the calculation of descriptive statistics and the statistical analysis, values as presented in the data listing will be used. Minimum and maximum will be presented to the same decimal precision as collected. Mean, median, and SD estimates will be presented to one decimal place

more than the precision of the data collected. CV will always be reported to 1 decimal place. Derived parameters will be reported using similar precision to those from which they were derived.

## 12 Study Subjects

The subsections in this section include specifications for reporting subject disposition and treatment/study discontinuations. Additionally, procedures for reporting protocol deviations are provided.

# 12.1 Disposition of Subjects and Discontinuations

The Investigator may withdraw a subject from the study based on following reasons:

- Withdrawal of subject's consent;
- Significant protocol violation, such as non-compliance with restriction regarding alcohol and drug use, and non-adherence to the fasting condition;
- Adverse events, as assessed by the Investigator to affect the subject safety or the outcome of the study endpoints;
- Difficulties with blood collection;
- Subject who vomits anytime during PK blood sampling will be excluded from the remainder of the study (including the rest of the periods if the adverse event occurred in the earlier ones). The subject will be advised to remain in the clinic for the rest of the confinement period for observation and so any safety related study procedures can be carried out;
- Subject reports adverse events of diarrhea (more than three episodes of loose stools) in any PK blood sampling period, which could render the plasma concentration-time profile unreliable;
- Subject is uncooperative during the study;
- Use of any ongoing or concomitant medication.

Subject may withdraw from the study at any time without any reason. Subjects who do not attend Study Check-In or withdraw during the study will be recorded in the Log Book of Non-Conformities Work. If the subject discontinues from the study at any time after taking the first dose of the study drug, the Case Report Form (CRF) would be completed accordingly and drug concentration will be analyzed. If a subject is discontinued early, all termination evaluations will be performed at the time of discontinuation. Details of reasons for premature withdrawal of subjects will be documented in the CSR.



#### 12.2 Protocol Deviations

# 12.2.1 Important Protocol Deviations

All protocol deviations will be listed in the CSR.

# 12.2.2 Reasons Leading to the Exclusion from an Analysis Set

All criteria/reasons leading to the exclusion of a subject from pharmacokinetic and statistical analyses will be summarized and listed in the CSR (see section 10.1).

# 13 Demographics and Other Baseline Characteristics

# 13.1 Demographics

Demographic characteristics will be reported (Table 1) using the following information from the Screening Visit CRF pages.

- Demographic characteristics
  - Gender: male, female
  - Race/Ethnic: Asian (Indonesia or other)
  - Age (years): summary statistics
  - Body weight
  - Body height
  - Body mass index (BMI)
  - Smoking status

Table 1 Demographic Data

| Demographic Characteristic | Statistics | Treatment Test Drug | Treatment Comparator Drug |
|---|---|---|---|
| | | (N =) | (N =) |
| Age (years) | Mean ± SD | $0.0 \pm 0.0$ | $0.0 \pm 0.0$ |
| | Range | 0 - 0 | 0 - 0 |
| Gender, n (%) | Male | 0 (0.0%) | 0 (0.0%) |
| | Female | 0 (0.0%) | 0 (0.0%) |
| Race, n (%) | Indonesian | 0 (0.0%) | 0 (0.0%) |
| | Other | 0 (0.0%) | 0 (0.0%) |
| Body weight (kg) | Mean ± SD | $0.00 \pm 0.00$ | $0.00 \pm 0.00$ |
| | Range | 0.0 - 0.0 | 0.0 - 0.0 |
| Body height (cm) | Mean ± SD | $0.00 \pm 0.00$ | $0.00 \pm 0.00$ |
| | Range | 0.0 - 0.0 | 0.0 - 0.0 |
| Body Mass Index | Mean ± SD | $0.000 \pm 0.000$ | $0.000 \pm 0.000$ |
| | Range | 0.0 - 0.0 | 0.0 - 0.0 |
| Smoke, n (%) | Non-smoker | 0 (0.0%) | 0 (0.0%) |
| | Smoke <10 cig./day | 0 (0.0%) | 0 (0.0%) |

# 13.2 Medical History

Medical history of all subjects will be recorded in the CRF and will not be presented in the CSR.

## 13.3 Other Baseline Characteristics

Vital signs measurements (listed in Table 10), clinical laboratory test results, ECG findings, and physical examination during Screening will be recorded in the CRF and reported in the CSR (Table 2).

Table 2 Clinical Laboratory Test and ECG of Subjects

| Parameter | Unit | | Normal Values | | | |
|---|---|---|---|---|---|---|
| | | (SUBJECT ID) | (SUBJECT ID) | (SUBJECT ID) | (SUBJECT ID) | |
| | | (INITIAL) | (INITIAL) | (INITIAL) | (INITIAL) | |
| | | (GENDER) | (GENDER) | (GENDER) | (GENDER) | |
| Screening Hematology Leucocyte Erythrocyte Hb Hematocrit Thrombocyte | $\begin{array}{c} x \ 10^{3}/\mu L \\ x \ 10^{6}/\mu L \\ g/dL \\ \frac{9}{6} \\ x \ 10^{3}/\mu L \end{array}$ | | | | | M:3.8 - 10.6 F: 3.6 - 11.0<br>M:4.4 - 5.9 F: 3.8 - 5.2<br>M:13.2 - 17.3 F: 11.7 - 15.5<br>M:40 - 52 F: 35 - 47<br>150 - 440 |
| Sero-immunology<br>HBsAg<br>Anti-HCV<br>Anti-HIV | | | | | | Neg.<br>Neg.<br>Neg. |
| Blood Chemistry Total bilirubin Direct bilirubin AST ALT AP Albumin Total protein Blood glucose Ureum Creatinine | mg/dL<br>mg/dL<br>IU/L<br>IU/L<br>g/dL<br>g/dL<br>mg/dL<br>mg/dL<br>mg/dL | | | | | <1.2 <0.50 M: <35 F: <31 M: <45 F:<34 M: 53 - 128 F: 42 - 98 3.5 - 5.2 6.4 - 8.3 <140 13 - 43 M: 0.67 - 1.17 F: 0.51 - 0.95 |
| Urinalysis Clarity Color Glucose Bilirubin Ketone Specific Gravity Blood pH Protein Urobilinogen Nitrite Leucocyte | EU/dL | | | | | Clear Yellow Neg. Neg. Neg. 1.015 - 1.025 Neg. 5 - 8 Neg. 0.2 - 1.0 Neg. Neg. |
| Sediment: - RBC - WBC - cast - epithel: squamous transitional tubular - crystal - bacteria | cells/HPF<br>cells/HPF | | | | | 0 - 2<br>0 - 5<br>Neg.<br>Neg./ Pos.<br>Neg./ Pos.<br>Neg./ Pos.<br>Neg. for male |



| Parameter | Unit | | Normal Values | | | |
|---|---|---|---|---|---|---|
| | | (SUBJECT ID) (SUBJECT ID) (SUBJECT ID) | | | | |
| | | (INITIAL) | (INITIAL) | (INITIAL) | (INITIAL) | |
| | | (GENDER) | (GENDER) | (GENDER) | (GENDER) | |
| Alcohol Test | | | | | | |
| Urine Drug Test - Barbiturates - Cocaine - Amphetamine - Cannabinoid - Morphine - Benzodiazepine Urine HCG Test | | | | | | Neg.<br>Neg.<br>Neg.<br>Neg. |
| ECG Conclusion | | | | | | Normal Sinus Rhythm |
| Period 1<br>Alcohol test | | | | | | Neg. |
| Urine Drug Test - Barbiturates - Cocaine - Amphetamine - Cannabinoid - Morphine - Benzodiazepine Urine HCG Test | | | | | | Neg.<br>Neg.<br>Neg.<br>Neg. |
| Period 2<br>Alcohol test | | | | | | Neg. |
| Urine Drug Test - Barbiturates - Cocaine - Amphetamine - Cannabinoid - Morphine - Benzodiazepine Urine HCG Test | | | | | | Neg.<br>Neg.<br>Neg.<br>Neg. |

<sup>\*</sup>deviate from normal values, but not clinically significant

#### 14 Previous or Concomitant Medications/Procedures

**Concomitant treatments** are medications, other than investigational product, which are taken by subjects any time during the study.

**Previous medications** are medications, other than investigational product, which started within 14 days before first drug administration.

All previous or concomitant medications, which were undertaken any time during study, will be summarized in the CRF. The Brand/Generic Name of the concomitant medications will be reported in the CRF.

 $<sup>^{\</sup>circ}$  lead to screen failure

# 15 Treatment Compliance and Exposure

This bioequivalence study is a single oral dose administration.

All dosing and treatment compliance, including the date and time of drug administration, will be recorded on "B2 Dosing" and "C2 Dosing" CRFs pages and will not be presented in the CSR.

# **Endpoint Evaluation**

### 16.1 Primary Endpoint Analyses

The primary endpoints are  $C_{max}$  and  $AUC_{0-t}$  for metformin concentration in plasma.

The statistical method for testing bioequivalence is ANOVA for 2-period, 2-sequence, 2-treatment cross-over comparing  $AUC_{0-t}$  and  $C_{max}$  after ln transformation of the original values.

Bioequivalence is concluded if the 90% confidence interval of the Test/Reference geometric means ratio is in the range of 80.00-125.00% for AUC<sub>0-t</sub> and C<sub>max</sub>. This acceptance criterion is according to the Guideline on the Investigation of Bioequivalence, EMA, London, 2010; ASEAN Guideline for the Conduct of Bioequivalence Study, Lao PDR, 2015; and Indonesian guidelines, *Pedoman Uji Bioekivalensi, Badan Pengawas Obat dan Makanan (BPOM)*, Jakarta, 2015, page 37-38.

Phoenix® WinNonlin (PPD ) will be used to perform the statistical analyses of AUC<sub>0-t</sub> and C<sub>max</sub> using analysis of variance (ANOVA) with the factors TREATMENT, PERIOD, SEQUENCE and SUBJECT(SEQUENCE) after transformation of the data to their natural logarithmic (ln) values. Mean treatment differences will be estimated using the ANOVA model above. 90% confidence intervals will be computed for the treatment differences based on the residual error term. Differences and CIs will result in ratios and corresponding CIs after back-transformation.

# 16.2 Secondary Endpoint Analyses

The secondary endpoints are  $t_{max}$ , AUC<sub>0-inf</sub> and  $t_{1/2}$  for metformin concentration in plasma.

The difference in  $t_{max}$  will be analyzed non-parametrically on the original data using Wilcoxon matched-pairs test.

The  $t_{1/2}$  difference will be analyzed using Student's paired t-test or Wilcoxon matched-pairs test depending whether the differences of the paired data were distributed normally or not (tested with *Kolmogorov-Smirnov*).

#### 16.3 Estimation of Individual PK Parameters

Pharmacokinetic parameters will be calculated using standard non-compartmental methods Phoenix® WinNonlin® version 8.0, or higher (PPD ) as defined below

| Symbol | Definition |
|---|---|
| AUC <sub>0-t</sub> | area under plasma concentration curve from administration to last observed concentration at time t |
| AUC <sub>0-inf</sub> | Area under plasma concentration from time zero (dosing time) extrapolated to infinite time. AUC <sub>0-inf</sub> will be calculated as AUC <sub>0-t</sub> + $C_t/k_e$ , where $C_t$ is the last observed plasma concentration; $k_e$ is the terminal elimination rate constant and will be determined by least-squares regression analysis during the terminal log-linear phase of the concentration–time curve |
| C <sub>max</sub> | Maximum observed plasma concentration |
| t <sub>1/2</sub> | Terminal phase half-life time. $t_{1/2} = \ln (2)/k_e$ |
| t <sub>max</sub> | The time to reach the maximum observed concentration (C <sub>max</sub> ) |

All concentration values below the quantification limit (BQL) will be set to zero for all pharmacokinetic and statistical calculations.

# 17 Safety Evaluation

In this study, safety will be assessed by qualified study personnel by evaluating reported adverse events, clinical laboratory test results, vital signs measurements, ECG findings, physical examination findings (including body weight and height measurements), and use of concomitant medication. Adverse events, laboratory tests and vital signs will be recorded in the CRF and tabulated in the CSR.

#### 17.1 Adverse Events

An adverse event is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. WHO-ART will be used as coding dictionary of adverse events. All adverse events will be listed.

The following summary tables will be presented for treatment emergent AEs:

- Summary of TEAEs by SOC, PT and treatment
- Summary of TEAEs by SOC, PT, intensity and treatment



• Summary of TEAEs by SOC, PT, causality and treatment

The denominator for the percentages in the summaries will be the number of subjects in the safety population for each treatment.

# 17.1.1 All Adverse Events

All of adverse events occurred during the study will be listed in the CSR (Table 3). An overview of all adverse events will be presented in Table 4. Adverse reaction (from test and comparator drug) would be categorized as unrelated, unlikely, possibly related, probably, and definite related based on literature data and pharmacokinetics profile (Table 5). All adverse events, regardless of severity, will be followed up and recorded by the investigator. All adverse events will be recorded in the CRF and tabulated in the CSR.



Table 3 List of Adverse Events Occurred

| | Listing All Adverse Events | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Period (I or II)<br>Treatment | Subject<br>No. | System Organ Class/<br>Preferred Term/<br>Reported Term | Serious<br>criteria | Start Date | End Date<br>(AE Duration) | Severity | Relationship<br>to IMP | Action taken with study treatment | Other action taken | Outcome | Comment |
| Period I Reference | | /<br>/<br> | No | yyyy-mm-dd,<br>hh:mm | yyyy-mm-dd,<br>hh mm<br>(dd,hh,mm) | | | | | | |
| Period 2 Test | | | | | | | | | | | |

Table 4 Overview of all Adverse Events (by Group and Overall)

| | Test Drug<br>(N=xx) | Comparator Drug (N=xx) | All (N=xx) |
|---|---|---|---|
| Subjects with any AE (%) | 0 (00.0%) | 0 (00.0%) | 0 (00.0%) |
| Number of all AEs | 0 | 0 | 0 |
| Number of treatment emergent AEs | 0 | 0 | 0 |
| Drug-related AEs | 0 | 0 | 0 |
| Serious AEs | 0 | 0 | 0 |
| Withdrawal due to AEs | 0 | 0 | 0 |

**Table 5** Adverse Events: Number Observed

| Adverse event | vent Mild | | Moderate | | | Severe | | | | Total | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Definite | Probably | Possibly | Unlikely | Unrelated | Definite | Probably | Possibly | Unlikely | Unrelated | Definite | Probably | Possibly | Unlikely | Unrelated | |
| Test Drug | | | | | | | | | | | | | | | | |
| SOC 1 | | | | | | | | | | | | | | | | |
| | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |
| SOC 2 | | | | | | | | | | | | | | | | |
| ••• | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |
| SOC 3 | | | | | | | | | | | | | | | | |
| ••• | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |
| Others | | | | | | | | | | | | | | | | |
| ••• | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |
| Comparator Drug | | | | | | | | | | | | | | | | |
| SOC 1 | | | | | | | | | | | | | | | | |
| ••• | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |
| SOC 2 | | | | | | | | | | | | | | | | |
| ••• | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |
| SOC 3 | | | | | | | | | | | | | | | | |
| ••• | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |
| Others | | | | | | | | | | | | | | | | |
| | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0.0%) |

# 17.1.2 Adverse Events Leading to Treatment Discontinuation

All adverse events leading to withdrawal of the subject will be recorded in the CRF and tabulated in the CSR (Table 6).

Table 6 Listing of Subjects Who Dropped Out from Study

| Treatment | Subjects<br>No. | Age<br>(yr) | Last PK Sampling (date and actual time) | Duration | Dose | Concomitant<br>Medication | Reason for<br>Discontinuation |
|---|---|---|---|---|---|---|---|
| | | | yyyy-mm-dd,<br>hh:mm | yyyy-mm-dd,<br>hh:mm<br>(dd,hh,mm) | | | |
| | | | | | | · | |

Test drug: Glucophage® XR (PT Merck Tbk, Indonesia) Comparator drug: Glucophage® XR (Merck Sante, France)

# 17.2 Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

#### 17.2.1 **Deaths**

All serious adverse events that may result in death will be recorded in the SAE form and attached to the CRF. The summary of death cases will be tabulated in the CSR (Table 7).

Table 7 Listing of Deaths During the Study

| Period<br>(Treatment) | Subject No. | Serious Adverse<br>Event | Date and Time of Death | Comments |
|---|---|---|---|---|
| Test drug: Glucophage® XR (PT Merck Tbk, Indonesia) | | | | |

Test drug: Glucophage® XR (PT Merck Tbk, Indonesia) Comparator drug: Glucophage® XR (Merck Sante, France)

#### 17.2.2 Serious Adverse Events

All serious adverse events will be recorded in the SAE form and attached to the CRF. The summary of serious adverse events will be tabulated in the CSR (Table 8).

**Table 8** Listing of Serious Adverse Events

| Period<br>(Treatment) | Subject<br>No. | Serious<br>Adverse<br>Event | Start Date<br>(yyyy,mm,dd,<br>hh:mm) | End Date<br>(yyyy,mm,dd,<br>hh:mm) | Intensity | Causality | Time of drug<br>Administration | Withdrawal/<br>Drop-out | Outcome<br>(observed<br>until FU<br>visit) |
|---|---|---|---|---|---|---|---|---|---|

Test drug: Glucophage® XR (PT Merck Tbk, Indonesia) Comparator drug: Glucophage® XR (Merck Sante, France)

# 17.3 Clinical Laboratory Evaluation

All clinical laboratory results will be recorded in the CRF and tabulated in the CSR. Baseline clinical laboratory test results will be presented alongside vital signs measurements, ECG findings, and physical examination performed during Screening in Table 9 (see Section 13.3). Clinical laboratory test results and other characteristics during Follow-Up Visit will be presented as shown (Table 9).



Table 9 Clinical Laboratory Test and ECG of Subjects During Follow-Up Visit

| Parameter | Unit | | Normal Values | | | |
|---|---|---|---|---|---|---|
| | | | (Init | tials) | | |
| | | (SUBJECT ID) | (SUBJECT ID) | (SUBJECT ID) | (SUBJECT ID) | |
| | | (INITIAL) | (INITIAL) | (INITIAL) | (INITIAL) | |
| | | (GENDER) | (GENDER) | (GENDER) | (GENDER) | |
| Hematology Leucocyte Erythrocyte Hb Hematocrit Thrombocyte Blood Chemistry | x 10 <sup>3</sup> /μL<br>x 10 <sup>6</sup> /μL<br>g/dL<br>%<br>x 10 <sup>3</sup> /μL | | | | | M :3.8 - 10.6 F: 3.6 - 11.0<br>M :4.4 - 5.9 F: 3.8 - 5.2<br>M:13.2 - 17.3 F: 11.7 - 15.5<br>M :40 - 52 F: 35 - 47<br>150 - 440 |
| Total bilirubin Direct bilirubin AST ALT AP Albumin Total protein Blood glucose Ureum Creatinine | mg/dL<br>mg/dL<br>IU/L<br>IU/L<br>IU/L<br>g/dL<br>g/dL<br>mg/dL<br>mg/dL<br>mg/dL | | | | | <1.2<br><0.50<br>M: <35 F: <31<br>M: <45 F:<34<br>M: 53 - 128 F: 42 - 98<br>3.5 - 5.2<br>6.4 - 8.3<br><140<br>13 - 43<br>M: 0.67 - 1.17 F: 0.51 - 0.95 |
| Urinalysis Clarity Color Glucose Bilirubin Ketone Specific Gravity Blood pH Protein Urobilinogen Nitrite Leucocyte Sediment: | EU/dL | | | | | Clear Yellow Neg. Neg. Neg. 1.015 - 1.025 Neg. 5 - 8 Neg. 0.2 - 1.0 Neg. Neg. |
| - RBC - WBC - cast - epithel: squamous transitional tubular - crystal - bacteria ECG Conclusion | cells/HPF<br>cells/HPF | | | | | 0 - 2 0 - 5 Neg. Neg./ Pos. Neg./ Pos. Neg./ Pos. Neg./ Pos. Neg./ Pos. Neg. for male Normal Sinus Rhythm |

<sup>\*</sup>deviate from normal values, not clinically significant \*\* clinically relevant deviation for repeated measurement please refer to Table 10 unscheduled measurements



# 17.4 Vital Signs

Vital signs will be recorded in the CRF and tabulated in the CSR (Table 10).

**Table 10** Vital Signs Monitoring

| Subject No. | Period | Vital Signs | Screening | Day 1 | | Day 2 | | Follow | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Pre-dose | 2h | 4h | 6h | 8h | 12h | 24h | 32h | -Up |
| S1 | 1 | Systolic BP (mmHg) | | | | | | | | | | |
| | | Diastolic BP (mmHg) | | | | | | | | | | |
| | | Pulse rate (beats/min) | | | | | | | | | | |
| | | Respiratory rate (times/min) | | | | | | | | | | |
| | 2 | Systolic BP (mmHg) | | | | | | | | | | |
| | | Diastolic BP (mmHg) | | | | | | | | | | |
| | | Pulse rate (beats/min) | | | | | | | | | | |
| | | Respiratory rate (times/min) | | | | | | | | | | |
| S2 | 1 | Systolic BP (mmHg) | | | | | | | | | | |
| | | Diastolic BP (mmHg) | | | | | | | | | | |
| | | Pulse rate (beats/min) | | | | | | | | | | |
| | | Respiratory rate (times/min) | | | | | | | | | | |
| | 2 | Systolic BP (mmHg) | | | | | | | | | | |
| | | Diastolic BP (mmHg) | | | | | | | | | | |
| | | Pulse rate (beats/min) | | | | | | | | | | |
| | | Respiratory rate (times/min) | | | | | | | | | | |

Unscheduled measurements will be listed in Table 11.

**Table 11** Unscheduled Measurement

| Subject No. | Parameter | Result | Outcome |
|-------------|-----------|--------|---------|

# 17.5 Other Safety or Tolerability Evaluations

Not applicable

#### 18 Benefit Risk Assessment

Not applicable.

#### 19 References

Badan Pengawas Obat dan Makanan Republik Indonesia. Pedoman Uji Bioekivalensi. Jakarta: BPOM; 2015.

Chow SC, Wang H. On Sample Size Calculation in Bioequivalence Trials. Journal of Pharmacokinetics and Pharmacodynamics. 2001; 28(2): 155-169.

Dixon W.J., Massey F. J. Introduction to Statistical Analysis. McGraw-Hill. New York. 1969. p 449.

European Medicines Agency. Guideline on the Investigation of Bioequivalence. London: European Medicines Agency; 2010.

Food and Drug Administration. Bioanalytical Method Validation Guidance for Industry. May 2018.

ICH E3 Expert Working Group. Structure and Content of Clinical Study Reports. ICH Harmonised Tripartite Guideline; 1995.

ICH E9 Expert Working Group. Statistical Principles for Clinical Trials. ICH Harmonised Tripartite Guideline; 1998.